CLINICAL TRIAL: NCT04522479
Title: Comparison of Efficacy and Safety of Controlled Hyperstimulation of Prolonged Protocol in Early Follicular or Mid Luteal Phase: a Single Center, Randomized, Controlled Trial
Brief Title: Prolonged Protocol of Early Follicular or Mid Luteal Phase
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2019-07-115
Record Dates: First submitted 2020-07-17; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: IVF
Keywords: prolonged protocol; In vitro fertilization (IVF); Intracytoplasmic sperm injection (ICSI); single blastocyst transfer

STUDY DESIGN:
Intervention Model Description: The early follicular and mid luteal prolonged regimens were randomly enrolled in a ratio of 1 to 1
Who Masked: Investigator
Masking Description: Statistician blindness
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prolonged protocol of early follicular phase (No Intervention): Inject a full dose of GnRH-a in 1st-3rd day of menstruation (leuprorelin acetate, injection, 3.75mg), the level of E2, P, LH in peripheral blood and the number of follicles in bilateral internal ovarian sinuses were monitored 32-38 days after the depression. If the pituitary desensitization was achieved, Gn (recombinant human follicle stimulating hormone or urofollicle stimulating hormone, injection, 75-300iu) was used for contralled hyperstimulation, when the diameter of 2 follicles was ≥ 18mm，hCG (human chorionic gonadotropin, injection, 4000-10000IU) was used to trigger and retrieve the oocyte. Selective single blastocyst transplantation was performed on the 4th-6th day after the oocyte retrieved. β-hCG was detected on the 12th day after embryo transplantation, and pregnancy or not was judged. If patients get pregnancy, follow-up was continued until the 42nd day after baby delivery.
- prolonged protocol of middle luteal phase (Experimental): Inject a full dose of GnRH-a in 21st-23rd day of menstruation (leuprorelin acetate, injection, 3.75mg), the level of E2, P, LH in peripheral blood and the number of follicles in bilateral internal ovarian sinuses were monitored 32-38 days after the depression. If the pituitary desensitization was achieved, Gn (recombinant human follicle stimulating hormone or urofollicle stimulating hormone, injection, 75-300iu) was used for contralled hyperstimulation, when the diameter of 2 follicles was ≥ 18mm，hCG (human chorionic gonadotropin, injection, 4000-10000IU) was used to trigger and retrieve the oocyte. Selective single blastocyst transplantation was performed on the 4th-6th day after the oocyte retrieved. β-hCG was detected on the 12th day after embryo transplantation, and pregnancy or not was judged. If patients get pregnancy, follow-up was continued until the 42nd day after baby delivery.
  Interventions: Other: Change the injection time of long acting GnRH-a

INTERVENTIONS:
Other: Change the injection time of long acting GnRH-a — The whole dose of long acting GnRH-a drug was changed to be injected on day 21st-23rd day of menstruation
  Arms: prolonged protocol of middle luteal phase

SUMMARY:
Due to the injection of gonadotropin releasing hormone agonist (GnRH-a) before controlled ovarian hyperstimulation (COH), the scheme of prolonged early follicular period protocol has obvious advantages in achieving ideal egg number, increasing endometrial receptivity to embryo transfer, inhibiting endogenous luteinizing hormone (LH) peak and reducing cycle cancellation rate. The full dose of long acting GnRH-a was also applied before COH in the mid luteal Hypergrowth program, and the mechanism of its lowering tone was similar. But whether the clinical and perinatal outcome of early follicular hyperlengthening is as effective as that of mid luteal hyperlengthening has not been reported at home and abroad. Moreover, there is a lack of prospective randomized controlled studies.

DETAILED DESCRIPTION:
One injection of 3.75mg GnRHa was injected on the 1st-3rd or 21st-23rd day of menstruation. The level of estradiol (E2), progesterone (P), luteinizing hormone (LH) in peripheral blood and the number of follicles in bilateral ovarian internal sinuses were monitored on the 32nd-38th day after pituitary hyporegulation.Gonadotropin (Gn) will be given after pituitary desensitization. When the diameter of at least two follicles ≥ 18mm or more than three follicles ≥ 17mm, the trigger of human chorionic gonadotropin (hCG) will be given and oocyte will be retrieved. The selective fresh single blastocyst transplantation will be carried out on the 4th-6th day after oocyte retrieval. HCG test at 12nd day after transplatation. Follow-up investigation will given during the pregnancy and perinatal period.

ELIGIBILITY:
Inclusion Criteria:

1. Tubal factor infertility;
2. polycystic ovary (PCO) or polycystic ovary syndrome (PCOS) patients;
3. Patients of mild to moderate endometriosis；
4. Oligoasthenospermia in male；
5. More than 5 antral follicle count (AFC) on both ovaries；
6. Unexplained infertility: there is a history of no contraception and pregnancy for more than 1 year, no clear cause of infertility such as ovulation, fallopian tube, endometrium and male factors is found, or the above factors return to normal after treatment.

Exclusion Criteria:

1. History of adverse pregnancy and childbirth；
2. Unilateral ovariectomy；
3. Uterine malformation, intrauterine adhesion, submucous myoma；
4. Chromosomal abnormality of both husband and wife；
5. Patients with contraindications of assisted reproductive technology or pregnancy: such as uncontrolled diabetes mellitus, undiagnosed liver and kidney dysfunction, history of deep vein thrombosis, history of pulmonary embolism, history of cerebrovascular accident, uncontrolled hypertension, heart disease, suspected cervical cancer, endometrial cancer, breast cancer or previous history, undetermined vaginal bleeding;
6. Unable to be regularly follow up；
7. Participating in other clinical trials；
8. No fresh single blastocyst transfer.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1150 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2023-05-13 (Estimated); Study Completion 2024-05-13 (Estimated)

PRIMARY OUTCOMES:
live birth rate | live birth of more than 28 pregnancy weeks
  live birth rate per transplantation cycle

SECONDARY OUTCOMES:
clinical pregnancy rate | fetal heart beat confirmed by transvaginal ultrasound 26-35 days after embryo transplantation
  fetal heart beat confirmed by transvaginal ultrasound
good quality blastocyst rate | The ratio of good quality blastocysts above 4BB degree 4-6 days after oocyte collection
  formation rate of more than 4BB Blastocyst
Incidence rate of early on-set severe ovarian hyperstimulation syndrome (OHSS) | Severe ovarian hyperstimulation syndrome according to Golan standard within 7 days after ovum removal
  Severe ovarian hyperstimulation syndrome according to Golan standard
Early misscarage rate | Abortion before 12 pregnancy weeks
  Transvaginal sonography identified patients with abortion after clinical pregnancy
Perinatal complications | Incidence rate of mother and child complications from pregnancy to postpartum in 42 days
  Perinatal complications of mothers and fetus

CONTACTS AND LOCATIONS:
Overall Officials: Yingfen Ying, Principal Investigator — The 2nd Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT04522479/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT04522479/ICF_001.pdf